CLINICAL TRIAL: NCT03447912
Title: Smoke-free Air Coalitions in Georgia and Armenia: A Community Randomized Trial
Brief Title: Smoke-free Air Coalitions in Georgia and Armenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Michelle C. Kegler, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00097093; R01TW010664 (NIH)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Smoking
Keywords: Behavioral intervention; Social intervention; Public health; Smoking behavior
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: This is a matched-pairs community randomized controlled trial. 14 communities will receive the behavioral intervention and 14 will serve as control communities. Enrollment is on the community level rather than individual level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): Fourteen communities will be assigned to the intervention.
  Interventions: Behavioral: Intervention Condition
- Control Condition (No Intervention): The 14 communities assigned as controls will participate in the population-level survey and will be provided with a site-specific summary of findings but will not participate in any aspects of the intervention. To examine potential contamination in the control communities, a follow-up interview will be conducted with public health center leaders to assess any local coalition or grassroots actions regarding tobacco control that may have naturally occurred or be influenced by coalition activity in other communities.

INTERVENTIONS:
Behavioral: Intervention Condition — The intervention approach will be informed by the Community Coalition Action Theory (CCAT) developed by Butterfoss and Kegler. CCAT posits that coalitions form due to a threat, opportunity, or mandate. Public health center staff will form a coalition by recruiting partner organizations from civil society and other government sectors (e.g., health care, education), conduct situational assessment, and develop and implement action plans to promote the adoption and enforcement of smoke-free policies in public indoor and and outdoor spaces.
  Arms: Intervention Condition

SUMMARY:
This is a matched-pairs community randomized controlled trial (CRCT) to examine the impact of coalitions promoting smoke-free air policies on individual secondhand smoke exposure (SHSe).

This proposal will build the capacity of Georgia (GE) and Armenia (AM) researchers to conduct high-quality mixed methods tobacco research and test the Community Coalition Action Theory (CCAT) as a framework for impacting local community-driven policy change to inform such processes for the region more broadly. Researchers from the GE National Center for Disease Control (NCDC) and AM National Institute of Health (NIH) will collaborate with Emory to execute the proposed research, train tobacco control researchers within their organizations and partnering universities, and train practitioners within local communities to build local coalitions for tobacco control policy.

Twenty-eight communities (14 per country) will participate in the population-level tobacco survey at baseline and follow-up. Within each country, 7 communities will be randomized to the intervention condition and 7 to the control condition (14 communities per condition). In the intervention communities, public health center staff will form a coalition by recruiting partner organizations from civil society and other government sectors (e.g., health care, education), conduct situational assessment, and develop and implement action plans to promote the adoption and enforcement of smoke-free policies primarily in indoor and outdoor public places (e.g., worksites, hospitality). The GE NCDC and AM NIH will establish subcontracts with the local public health centers in the randomly selected communities to provide funding for local staff to develop local coalitions and to support program activities. The 14 communities assigned as controls will participate in the population-level survey and be provided with a site-specific summary of findings but will not participate in any aspects of the intervention. Additionally, to examine potential contamination in the control communities, a follow-up interview will be conducted with public health center leaders to assess any local coalition or grassroots actions regarding tobacco control that may have naturally occurred or be influenced by coalition activity in other communities.

DETAILED DESCRIPTION:
Public health efforts in low- and middle-income countries (LMICs) could be catalyzed by bolstering ways to optimally leverage local talents and resources, such as civil society. Developing effective models for aligning civil society and governmental public health at the local level in LMICs has the potential to impact a range of chronic diseases and risk factors, including tobacco use. Local coalitions have been a dominant strategy in tobacco control in the US, with well-documented success in establishing smoke-free policies specifically. However, this approach has not been widely leveraged or well-studied in LMICs or those with less democratic traditions than the US. Instead, in many LMICs, smoke-free policy progress is largely initiated at the national level. Parallel civil society movements at the local level may be needed to build support for and compliance with policies. Given their sociopolitical histories and high tobacco use and secondhand smoke exposure (SHSe) rates, Georgia (GE) and Armenia (AM) are two strategic settings for the proposed work. The smoking prevalence is 57.7% and 52.3% in men (6th and 11th highest in the world) and 5.7% and 1.5% in women, respectively. Moreover, previous findings indicate extremely high rates of SHSe. However, there is also documented high receptivity to public smoke-free policies despite high use rates.

In this matched-pairs community randomized controlled trial (CRCT), the impact of coalitions promoting smoke-free air policies on individual secondhand smoke exposure (SHSe) will be examined. The Emory team will lead the oversight of the research design and execution of all components of the research. This proposal will build the capacity of Georgia (GE) and Armenia (AM) researchers to conduct high-quality mixed methods tobacco research and test the Community Coalition Action Theory (CCAT) as a framework for impacting local community-driven policy change to inform such processes for the region more broadly. Researchers from the GE National Center for Disease Control (NCDC) and AM National Institute of Health (NIH) will collaborate with Emory to execute the proposed research, train tobacco control researchers within their organizations and partnering universities (Tbilisi State Medical University, American University of Armenia), and train practitioners within local communities to build local coalitions for tobacco control policy.

This study aims to:

1. conduct a matched-pair community randomized controlled trial in 28 municipalities in GE and AM to examine the impact of local coalitions promoting the adoption of smoke-free policies in public places, with the primary outcome of changes in SHSe over time;
2. assess how community context and coalition factors influence adoption of organizational and municipal smoke-free policies to provide an evidence-base for public health practice;
3. disseminate research findings regarding both the effectiveness and the process of establishing and maintaining coalitions, and consequently increasing smoke-free policies and reducing SHSe, to key stakeholders in GE and AM; and
4. capitalize on the proposed research and dissemination opportunities to build tobacco control research capacity within the GE NCDC, AM NIH, and partnering universities, as well as practice capacity within local public health centers and their civil society partners.

Twenty-eight communities (14 per country) will participate in the population-level tobacco survey at baseline and follow-up. Within each country, 7 communities will be randomized to the intervention condition and 7 to the control condition (14 communities per condition). In the intervention communities, public health center staff will form a coalition by recruiting partner organizations from civil society and other government sectors (e.g., health care, education), conduct situational assessment, and develop and implement action plans to promote the adoption and enforcement of smoke-free policies in primarily in indoor and outdoor public places (e.g., worksites, hospitality). The GE NCDC and AM NIH will establish subcontracts with the local public health centers in the randomly selected communities to provide funding for local staff to develop local coalitions and to support program activities. The 14 communities assigned as controls will participate in the population-level survey and be provided with a site-specific summary of findings but will not participate in any aspects of the intervention. Additionally, to examine potential contamination in the control communities, a follow-up interview will be conducted with public health center leaders to assess any local coalition or grassroots actions regarding tobacco control that may have naturally occurred or be influenced by coalition activity in other communities.

The GE NCDC and AM NIH will conduct cross-sectional population-level surveys in Year 1 (baseline) and in Years 4/5 (follow-up) in the intervention and control communities. A multi-stage, clustered sample design will be used to select 50 participants within each municipality. The most recent census data for each country and the respective municipalities will be used to establish the sampling frame.

ELIGIBILITY:
Community Level Inclusion Criteria:

* Population size ranging from approximately 6,000 to 90,000

Exclusion Criteria:

* Lack of interest of local health care center director

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2924 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kegler, DrPH, Principal Investigator — Emory University
Locations (2):
- National Institute of Health, Yerevan, Armenia
- National Center for Disease Control, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayrumyan V, Harutyunyan A, Torosyan A, Grigoryan L, Sargsyan Z, Bazarchyan A, Petrosyan V, Dekanosidze A, Sturua L, Kegler MC, Berg CJ. Tobacco-related risk perceptions, social influences and public smoke-free policies in relation to smoke-free home restrictions: findings from a baseline cross-sectional survey of Armenian and Georgian adults in a community randomised trial. BMJ Open. 2022 Feb 7;12(2):e055396. doi: 10.1136/bmjopen-2021-055396. PMID 35131832
- [Background] Berg CJ, Dekanosidze A, Hayrumyan V, LoParco CR, Torosyan A, Grigoryan L, Bazarchyan A, Haardorfer R, Kegler MC. Smoke-free home restrictions in Armenia and Georgia: motives, barriers and secondhand smoke reduction behaviors. Eur J Public Health. 2023 Oct 10;33(5):864-871. doi: 10.1093/eurpub/ckad129. PMID 37500602
- [Derived] Berg CJ, Haardorfer R, Torosyan A, Dekanosidze A, Grigoryan L, Sargsyan Z, Hayrumyan V, Sturua L, Topuridze M, Petrosyan V, Bazarchyan A, Kegler MC. Examining local smoke-free coalitions in Armenia and Georgia: context and outcomes of a matched-pairs community-randomised controlled trial. BMJ Glob Health. 2024 Feb 7;9(2):e013282. doi: 10.1136/bmjgh-2023-013282. PMID 38325896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were from communities in Tbilisi, Georgia and Yerevan, Armenia. Community member participation began October 1, 2018 and the follow-up assessments occurred in Spring and Summer of 2022 (approximately 44 months after the start of community member participation in the baseline surveys). Follow-up assessments were completed by June 30, 2022.
Pre-assignment Details: Fourteen communities delivered the study intervention and 14 continued as usual to serve as a control group. In this repeated cross-sectional study design, surveys were administered at baseline and follow-up (approximately 44 months after baseline) to community members. Individual community members were only assessed once, participating in either the baseline or follow-up time points.
Units Other Than Participants: communities
Groups:
- Intervention Condition: Community members in communities assigned to an intervention promoting the adoption and enforcement of smoke-free policies primarily in indoor and outdoor public places (e.g., worksites, hospitality) to reduce secondhand smoke exposure.
  The intervention approach was informed by the Community Coalition Action Theory (CCAT) developed by Butterfoss and Kegler. CCAT posits that coalitions form due to a threat, opportunity, or mandate. Public health center staff will form a coalition by recruiting partner organizations from civil society and other government sectors (e.g., health care, education), conduct situational assessment, and develop and implement action plans to promote the adoption and enforcement of smoke-free policies in indoor and outdoor public spaces.
- Control Condition: Community members in communities assigned to the control condition which participated in population-level surveys but did not participate in any aspects of the intervention.
Period: Overall Study
Arm/Group | Intervention Condition | Control Condition
Started | 1481; 14 communities | 1443; 14 communities
Community Members Who Completed the Baseline Survey | 732; 14 communities | 724; 14 communities
Community Members Who Completed the Follow-up Survey | 749; 14 communities | 719; 14 communities
Completed | 1481; 14 communities | 1443; 14 communities
Not Completed | 0; 0 communities | 0; 0 communities

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes community members who completed the baseline assessment.
Groups:
- Intervention Condition: Community members in communities assigned to an intervention promoting the adoption and enforcement of smoke-free policies primarily in indoor and outdoor public places (e.g., worksites, hospitality) to reduce secondhand smoke exposure.
- Total: Total of all reporting groups
Arm/Group | Intervention Condition | Control Condition | Total
Number analyzed (Participants) | 732 | 724 | 1456
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.52 (13.71) | 44.19 (13.22) | 43.35 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 429 | 452 | 881
  Male | 303 | 272 | 575
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 732 | 724 | 1456
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 732 | 724 | 1456
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Armenia | 351 | 354 | 705
  Georgia | 381 | 370 | 751

OUTCOME MEASURES:

1. Primary Outcome: Secondhand Smoke Exposure
Description: The frequency of secondhand smoke (SHS) exposure in the past 30 days was assessed by asking the respondent to report the number of days they were exposed to SHS.
Time Frame: Baseline, Follow-up (approximately 44 months post-baseline)
Population: This analysis includes community members who completed the Baseline or Follow-up assessments. Community members at each time point are distinct groups who participated in the study only once rather than at both time points.
Measure: Mean (Standard Deviation); unit: days with SHS exposure
Arm/Group | Intervention Condition | Control Condition
Number analyzed (Participants) | 1481 | 1443
days with SHS exposure
  Baseline: number analyzed (Participants) | 732 | 724
  Baseline | 11.70 (12.14) | 12.08 (12.35)
  Follow-up: number analyzed (Participants) | 749 | 719
  Follow-up | 10.86 (11.77) | 10.51 (11.92)

2. Secondary Outcome: Attitude Regarding Secondhand Smoke Exposure
Description: Attitudes regarding Secondhand Smoke Exposure (SHSe) were examined by assessing the degree to which the respondent believes that smoke causes illnesses. Participants were asked "Based on what you know or believe, does breathing other people's smoke cause serious illness in non-smokers?" Possible responses are 1 = "not at all", 2 = "a little", 3 = "somewhat", or 4 = "a lot".
Time Frame: Baseline, Follow-up (approximately 44 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Condition | Control Condition
Number analyzed (Participants) | 1481 | 1443
score on a scale
  Baseline: number analyzed (Participants) | 732 | 724
  Baseline | 2.53 (0.70) | 2.53 (0.68)
  Follow-up: number analyzed (Participants) | 749 | 719
  Follow-up | 3.44 (0.81) | 3.37 (0.82)

3. Secondary Outcome: Attitude Regarding Smoke-Free Environments
Description: To assess attitudes regarding smoke-free environments, respondents were asked whether they think smoking should or should not be allowed in places such as workplaces, indoor areas on school grounds, outdoor events, restaurants, and bars. Participants indicated how much the supported or opposed complete cigarette smoking bans on a 4-point scale where 1 = strongly oppose and 4 = strongly support.
Time Frame: Baseline, Follow-up (approximately 44 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Condition | Control Condition
Number analyzed (Participants) | 1481 | 1443
score on a scale
  Baseline - In restaurants, cafes, and cafeterias: number analyzed (Participants) | 732 | 724
  Baseline - In restaurants, cafes, and cafeterias | 3.36 (0.88) | 3.32 (1.02)
  Baseline - On the outdoor terrace of restaurants, cafes, and cafeterias: number analyzed (Participants) | 732 | 724
  Baseline - On the outdoor terrace of restaurants, cafes, and cafeterias | 2.39 (1.12) | 2.60 (1.21)
  Baseline - In bars, pubs, or nightclubs: number analyzed (Participants) | 732 | 724
  Baseline - In bars, pubs, or nightclubs | 3.05 (1.05) | 3.08 (1.17)
  Baseline - On the outdoor terrace of bars, pubs, or nightclubs: number analyzed (Participants) | 732 | 724
  Baseline - On the outdoor terrace of bars, pubs, or nightclubs | 2.33 (1.14) | 2.49 (1.24)
  Baseline - Indoor common areas of apartment or condominium complexes (hallways, lobbies, stairwells): number analyzed (Participants) | 732 | 724
  Baseline - Indoor common areas of apartment or condominium complexes (hallways, lobbies, stairwells) | 3.26 (0.96) | 3.21 (1.05)
  Baseline - Outdoor common areas of apartment or condominium complexes (playgrounds, park benches): number analyzed (Participants) | 732 | 724
  Baseline - Outdoor common areas of apartment or condominium complexes (playgrounds, park benches) | 3.10 (0.98) | 3.04 (1.07)
  Baseline - Within individual apartment or condo units within a complex: number analyzed (Participants) | 732 | 724
  Baseline - Within individual apartment or condo units within a complex | 3.17 (1.00) | 3.06 (1.14)
  Baseline - Private vehicles when children under age 18 are present: number analyzed (Participants) | 732 | 724
  Baseline - Private vehicles when children under age 18 are present | 3.84 (0.47) | 3.77 (0.61)
  Baseline - Parks and beaches: number analyzed (Participants) | 732 | 724
  Baseline - Parks and beaches | 2.93 (1.04) | 2.91 (1.09)
  Baseline - Other public outdoor areas, such as open stadiums: number analyzed (Participants) | 732 | 724
  Baseline - Other public outdoor areas, such as open stadiums | 2.86 (1.11) | 2.77 (1.18)
  Follow-up - In restaurants, cafes, and cafeterias: number analyzed (Participants) | 749 | 719
  Follow-up - In restaurants, cafes, and cafeterias | 3.36 (0.98) | 3.33 (1.00)
  Follow-up - On the outdoor terrace of restaurants, cafes, and cafeterias: number analyzed (Participants) | 749 | 719
  Follow-up - On the outdoor terrace of restaurants, cafes, and cafeterias | 2.59 (1.15) | 2.49 (1.12)
  Follow-up - In bars, pubs, or nightclubs: number analyzed (Participants) | 749 | 719
  Follow-up - In bars, pubs, or nightclubs | 3.26 (1.04) | 3.32 (1.00)
  Follow-up - On the outdoor terrace of bars, pubs, or nightclubs: number analyzed (Participants) | 749 | 719
  Follow-up - On the outdoor terrace of bars, pubs, or nightclubs | 2.59 (1.16) | 2.49 (1.12)
  Follow-up -Indoor common areas of apartment or condominium complexes (hallways, lobbies, stairwells): number analyzed (Participants) | 749 | 719
  Follow-up -Indoor common areas of apartment or condominium complexes (hallways, lobbies, stairwells) | 3.24 (1.01) | 3.17 (1.04)
  Follow-up - Outdoor common areas of apartment or condominium complexes (playgrounds, park benches): number analyzed (Participants) | 749 | 719
  Follow-up - Outdoor common areas of apartment or condominium complexes (playgrounds, park benches) | 2.97 (1.10) | 2.92 (1.08)
  Follow-up - Within individual apartment or condo units within a complex: number analyzed (Participants) | 749 | 719
  Follow-up - Within individual apartment or condo units within a complex | 3.06 (1.14) | 2.96 (1.20)
  Follow-up - Private vehicles when children under age 18 are present: number analyzed (Participants) | 749 | 719
  Follow-up - Private vehicles when children under age 18 are present | 3.62 (0.79) | 3.62 (0.80)
  Follow-up - Parks and beaches: number analyzed (Participants) | 749 | 719
  Follow-up - Parks and beaches | 2.74 (1.08) | 2.64 (1.07)
  Follow-up - Other public outdoor areas, such as open stadiums: number analyzed (Participants) | 749 | 719
  Follow-up - Other public outdoor areas, such as open stadiums | 2.82 (1.09) | 2.68 (1.08)

4. Secondary Outcome: Count of Participants Agreeing With Certain Home Policies
Description: Smoke-free home policies at baseline and follow-up were assessed by asking about rules about smoking inside of the participant's home. Possible responses included: smoking is allowed, smoking is not allowed but there are exceptions, smoking is never allowed, or there are no rules about smoking in the home.
Time Frame: Baseline, Follow-up (approximately 44 months post-baseline)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Condition | Control Condition
Number analyzed (Participants) | 1481 | 1443
Participants
  Baseline: number analyzed (Participants) | 732 | 724
  Baseline: Smoking is allowed | 91 | 110
  Baseline: Smoking is not allowed but there are exceptions | 209 | 177
  Baseline: Smoking is never allowed | 298 | 263
  Baseline: There are no rules about smoking in the home | 131 | 172
  Baseline: No response | 3 | 2
  Follow-up: number analyzed (Participants) | 749 | 719
  Follow-up: Smoking is allowed | 95 | 90
  Follow-up: Smoking is not allowed but there are exceptions | 147 | 136
  Follow-up: Smoking is never allowed | 418 | 369
  Follow-up: There are no rules about smoking in the home | 88 | 124
  Follow-up: No response | 1 | 0

5. Secondary Outcome: Count of Participants With Certain Workplace Policies
Description: Among participants employed in a workplace with an indoor setting, workplace policies at baseline and follow-up were measured by asking, "Which of the following best describes the indoor smoking policy where you work? Smoking is allowed anywhere, smoking is allowed only in some indoor areas, smoking is not allowed in any indoor areas, or there is no policy."
Time Frame: Baseline, Follow-up (approximately 44 months post-baseline)
Population: This analysis includes community members who work outside of the home in a workplace with an indoor setting and who completed the Baseline or Follow-up assessments. Community members at each time point are distinct groups who participated in the study only once rather than at both time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Condition | Control Condition
Number analyzed (Participants) | 682 | 600
Participants
  Baseline: number analyzed (Participants) | 340 | 307
  Baseline: Smoking is allowed anywhere | 32 | 38
  Baseline: Smoking is allowed only in some indoor areas | 51 | 28
  Baseline: Smoking is not allowed in any indoor areas | 217 | 173
  Baseline: There is no policy | 40 | 68
  Follow-up: number analyzed (Participants) | 342 | 293
  Follow-up: Smoking is allowed anywhere | 9 | 7
  Follow-up: Smoking is allowed only in some indoor areas | 46 | 42
  Follow-up: Smoking is not allowed in any indoor areas | 266 | 233
  Follow-up: There is no policy | 21 | 11

6. Secondary Outcome: Enforcement of Smoke-Free Policies
Description: Changes in enforcement of smoke-free policies in various settings will be measured by asking, "In the past 7 days, how many times have you seen someone using tobacco in a location where it is prohibited?"
Time Frame: Baseline, Follow-up (approximately 44 months post-baseline)
Population: This item was not administered at either study time point.
Arm/Group | Intervention Condition | Control Condition
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Secondhand Smoke Exposure in Various Locations
Description: The frequency of secondhand smoke (SHS) exposure in the past 30 days will be assessed by asking the respondent to report the number of days they were exposed to SHS in the home, in vehicles, at work, in indoor public places, and in outdoor public places. The frequency of exposures is evaluated as the number of days in the past 30 days the participant was exposed to SHS in the home, in vehicles, at work, in indoor public places, and in outdoor public places
Time Frame: Baseline, Follow-up (approximately 44 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days with SHS exposure
Arm/Group | Intervention Condition | Control Condition
Number analyzed (Participants) | 1481 | 1443
days with SHS exposure
  Baseline - Exposure in the home: number analyzed (Participants) | 732 | 724
  Baseline - Exposure in the home | 6.83 (11.48) | 7.18 (11.53)
  Baseline - Exposure in vehicles: number analyzed (Participants) | 732 | 724
  Baseline - Exposure in vehicles | 3.87 (8.15) | 3.93 (8.36)
  Baseline - Exposure in indoor work areas: number analyzed (Participants) | 732 | 724
  Baseline - Exposure in indoor work areas | 4.16 (8.66) | 4.44 (8.85)
  Baseline - Exposure in indoor public areas: number analyzed (Participants) | 732 | 724
  Baseline - Exposure in indoor public areas | 1.74 (4.71) | 2.00 (5.17)
  Baseline - Exposure in outdoor public areas: number analyzed (Participants) | 732 | 724
  Baseline - Exposure in outdoor public areas | 5.34 (8.86) | 4.83 (8.79)
  Follow-up - Exposure in the home: number analyzed (Participants) | 749 | 719
  Follow-up - Exposure in the home | 4.88 (9.83) | 4.72 (9.83)
  Follow-up - Exposure in vehicles: number analyzed (Participants) | 749 | 719
  Follow-up - Exposure in vehicles | 4.43 (8.27) | 4.74 (9.27)
  Follow-up - Exposure in indoor work areas: number analyzed (Participants) | 749 | 719
  Follow-up - Exposure in indoor work areas | 2.91 (7.70) | 3.06 (7.68)
  Follow-up - Exposure in indoor public areas: number analyzed (Participants) | 749 | 719
  Follow-up - Exposure in indoor public areas | 1.66 (5.21) | 1.15 (3.89)
  Follow-up - Exposure in outdoor public areas: number analyzed (Participants) | 749 | 719
  Follow-up - Exposure in outdoor public areas | 6.78 (9.68) | 6.49 (9.02)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected while community member participants were completing the Baseline or Follow-up survey (approximately 44 months post-baseline), which was completed within one hour on their single day of study participation.
Arm/Group | Intervention Condition | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/1481 | 0/1443
Serious Adverse Events (participants affected / at risk) | 0/1481 | 0/1443
Other Adverse Events (participants affected / at risk) | 0/1481 | 0/1443

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT03447912/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03447912/ICF_002.pdf